CLINICAL TRIAL: NCT02900235
Title: An Open-label, Mass Balance Study to Investigate the Absorption, Metabolism and Excretion of [14C]-MT-3995 After a Single Oral Dose to Healthy Male Subjects
Brief Title: Mass Balance Study of MT-3995
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MT-3995-E11
Record Dates: First submitted 2016-08-17; First posted 2016-09-14 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: Healthy
MeSH Terms: interventions — apararenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MT-3995 (Experimental): [14C]-MT-3995 after a single oral dose
  Interventions: Drug: MT-3995

INTERVENTIONS:
Drug: MT-3995

SUMMARY:
The purpose of this study is to investigate the absorption, metabolism and excretion of MT-3995 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent to participate in the study
* Caucasian male aged at least 35 years at Screening
* Healthy and free from clinically significant illness or disease at Screening and Day-1
* A body weight of 60 to 110 kg at Screening and Day-1
* Vital signs within the following ranges at Screening, Day-1 and Pre-dose:

  * Body temperature : 35.0°C to 37.5°C
  * Systolic blood pressure: 90 to 140 mmHg
  * Diastolic blood pressure: 50 to 90 mmHg
* Regular daily bowel movements

Exclusion Criteria:

* Presence or history of severe adverse reaction or allergy to any medicinal product
* Participation in more than three clinical studies of an Investigational Medicinal Product (IMP) in the previous year or participated in a clinical study of any IMP within 12 weeks or five half-lives
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardise the subject in case of participation in the study. The Investigator should be guided by evidence of any of the following:

  * History of inflammatory bowel syndrome, gastritis, ulcers, gastrointestinal or rectal bleeding considered clinically significant by the Investigator
  * History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy or bowel resection
  * History or clinical evidence of pancreatic injury or pancreatitis

Min Age: 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Total radioactivity in urine and faeces | up to 99 days
Maximum observed plasma concentration [Cmax] | up to 99 days
Time at which Cmax occurs [tmax] | up to 99 days
Area under the plasma concentration-time curve from time zero to the last measurable concentration [AUC0-t] | up to 99 days
Area under the plasma concentration-time curve from time zero to infinity [AUC0-∞] | up to 99 days
Apparent terminal elimination half-life [t1/2] | up to 99 days
Terminal elimination rate constant [Kel] | up to 99 days

SECONDARY OUTCOMES:
Safety and tolerability as measured by adverse events (AEs) | up to 99 days
Safety and tolerability as measured by vital signs | up to 99 days

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (1):
- Investigational center, City Name, United Kingdom